CLINICAL TRIAL: NCT03359824
Title: Brown Adipose Tissue Activation: Effect of Exercise Training and Irisin
Acronym: EXEBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Pirjo Nuutila, MD., Ph.D., Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EXEBAT
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Physical Activity
Keywords: exercise, brown adipose tissue
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Other): Arm: Exercise: Combination of moderate intensity continuous training, high intensity interval training and endurance training 5 times per week for a total of 6 weeks. Out of 5 sessions three were supervised by trainer and two sessions were performed by subjects on their own.The duration of the exercise was increased progressively. The first two weeks was 30 minutes that increased to 45 minutes in the third and fourth week. It was 60 minutes for the last two weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
This study investigates the brown adipose tissue (BAT) activation and metabolism using positron emission tomography (PET) imaging before and after exercise training intervention at fasting state under normal room temperature and during cold stimulation.The investigators hypothesize that BAT glucose uptake is increased after exercise and BAT becomes metabolically more active.

Understanding the mechanisms of BAT activation and the role of exercise in humans is crucial to combat epidemic of obesity and diabetes.

DETAILED DESCRIPTION:
Exercise training has been suggested to activate and recruit human BAT through the activation of sympathetic nervous system and contracting skeletal muscles by the release of myokines such as lactate and irisin that signal WAT to induce expression of beige adipocytes. It has been also suggested that exercise training could enhance the metabolism of already existed functional BAT by increasing uncoupling protein-1 (UCP-1) gene transcription, mitochondrial biogenesis and hyperplasia. This is of clinical relevance because brown fat activation has been found to improve metabolic factors linked to obesity and diabetes.

In this study the investigators use a PET radiotracer 2-[18F] flouro-2-deoxy-D-glucose (FDG) to quantify the glucose uptake in BAT, whie adipose tissue and the muscle.The participants are scanned thrice at fast in this study once at room temperature, second at cold exposure and third after six weeks of exercise at cold exposure. This study will provide an insight about the role of exercise in activation of BAT metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy sedentary volunteer

  1. BMI 20-25 kg/m2
  2. Age: 18-45 years
  3. No chronic diseases

Exclusion Criteria:

1. BMI < 20 kg/m2 or BMI > 25 kg/m2
2. Mental disorder or poor compliance
3. Eating disorder or excessive use of alcohol or tobacco smoking
4. Any chronic disease
5. Past dose of radiation
6. Presence of any ferromagnetic objects that would make MR imaging contraindicated
7. Physically disability which rule out the physical fitness tests or participation in the exercise training intervention
8. Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2015-05-27 (Actual); Study Completion 2015-05-27 (Actual)

PRIMARY OUTCOMES:
Cold-induced glucose uptake in BAT after exercise | Within one study day
  Glucose uptake of brown adipose tissue acquired with PET under cold exposure after exercise intervention. PET imaging is used to quantify glucose uptake in tissues

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, MD, PhD, Principal Investigator — Turku UH

IPD SHARING:
Plan to Share IPD: No